CLINICAL TRIAL: NCT01006148
Title: Comparison of Allogenix Plus Demineralized Bone Matrix and Autogenous Bone Dust Versus Autogenous Bone Dust Alone in Ossification of Small Calvarial Defects, a Pilot Study.
Brief Title: Comparison of a Bone Product to Bone Dust in Ossification of Small Calvarial Defects.
Acronym: DBM
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: problems obtaining the investigational agent, Allogenix(TM) Plus
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 1146218
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Metopic Craniosynostosis
Keywords: Metopic Craniosynostosis
MeSH Terms: conditions — Trigonocephaly, Nonsyndromic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bone substitute (Experimental): Enrollees will receive Allogenix Plus(TM), a demineralized bone matrix, to fill in calvarial gaps after cranial vault remodeling and fronto-orbital advancement.
  Interventions: Biological: Allogenix Plus

INTERVENTIONS:
Biological: Allogenix Plus — It is a demineralized bone matrix obtained using cortical or cancellous allograft bone that is treated to remove surface lipids and then dehydrated with ethanol and ethyl esther. It is further processed leaving behind proteins, bone growth factors, and collagen. It is combined with lecithin a which is resistant to breakdown by body fluids. It contains Pro Osteon Implant 500R a naturally derived material made from a non-decorative form of coral, which is subject to a patented thermal process, which converts the coral to hydroxyapatite.

SUMMARY:
In this study we want to compare the effectiveness of a bone substitute (Allogenix Plus, a product derived from a dead human being that has chosen to donate it prior to dying) and bone dust from the patient's own bone pieces, versus bone dust alone in filling in the gaps that sometimes occur after surgery for craniosynostosis . We will compare the percent of defect filled at 1 year in 5 patients 18 months or older with metopic craniosynostosis that received the bone substitute plus their bone dust with 5 previously operated patients with similar characteristics that received bone dust alone to fill in the gaps. The bone substitute that we are using will be provided at no cost by the company Biomet Microfixation. The bone substitute Allogenix Plus undergoes extensive screening for infectious diseases as well as processing to prevent a rejection. The product will be applied during standard surgery to 5 patients with metopic craniosynostosis of 18 months or older with skull defects no larger than 25 cm2, so it does not require any additional surgeries. Aside from the placement of this bone substitute the patient will proceed to receive the standard of care which includes a pre-operative CT scan, immediate post-operative CT scan, and 1 year post-operative CT scan of the Head. We will review these scans and look at percent of bony growth in the bone substitute plus bone dust group . We will also see the patients in clinic, during standard of care follow-up visits at 1 week, 3 weeks, 6 weeks, 12 weeks, 6 months, and 1 year post-operatively. During clinic visits we will monitor the patient closely for any potential side effects of the bone substitute as well as complications of the surgery. We will then review the charts of 5 patients 18 months or older that have undergone surgery for metopic craniosynostosis until 5 patients with similar characteristics and defect size have been obtained. We will compare their post-operative CT scans and pictures and we will look at bone growth, bone resorption, bone gaps present, and need for secondary surgeries.

DETAILED DESCRIPTION:
The skull is made of multiple bones that are separated from each other at the time of birth through sutures (joints). These sutures (open spaces) allow for growth of the brain resulting in growth of the skull bones. These sutures close at different stages of life, the metopic suture is the earliest one to close at 2 years old and the latest at 26 years old. If these sutures (open spaces) close prematurely the patient develops craniosynostosis. This will result in lack of growth of the skull perpendicular to the suture line and increased growth parallel to the suture. There are different degrees of craniosynostosis that will result in anything from a slight ridge along the suture line to abnormal head shape causing constriction of the brain, developmental delays, and elevated intracranial pressure. Patients with significant abnormal head shape or patients showing any developmental delay will undergo surgical intervention. The surgery is called Cranial Vault Remodeling and it consists of opening the scalp to access the skull bones involved, then removing the bones from the underlying brain, reshaping and expanding the bone, and placing them back to protect the brain. The skull bones are held together with absorbable plates. Because the skull bones are expanded to allow for adequate brain growth there are gaps that are left without any bone. Some of these gaps are filled in with the left over small bony pieces. Other gaps are filled in with even smaller pieces of left over bone that is placed in a saw mill to form bone dust. Often, the amount of bone dust and bone pieces is not enough to fill in all the gaps. When the gaps are left unfilled it usually takes longer for these areas to be filled by the patient's own bone. This means that the brain underneath these gaps is left unprotected until they are covered with bone. At times, primarily in children 18 months or older, we find that these gaps are never fully filled requiring the child to undergo a second surgery in which bone is taken either from the ribs or the skull to fill in these gaps. Specific Aims: 1) Evaluate the efficacy of the bone substitute Allogenix Plus in ossification of small cranial defects in patients with metopic craniosynostosis forms exist. These are derived from cadaver graft material that have been determined eligible for transplantation by a qualified tissue bank medical director and communicable disease testing has been performed by a laboratory certified under CLIA. Allogenix Plus is a demineralized bone matrix obtained using cortical or cancellous allograft bone that is treated to remove surface lipids and then dehydrated with ethanol and ethyl esther. The bone is further processed with hyaluronic acid to remove acid-soluble proteins in the bone, leaving behind other proteins, bone growth factors, and collagen. The demineralized bone matrix is then combined with lecithin a non-toxic lipid carrier derived from soybeans that is resistant to breakdown by body fluids. It also contains an additional synthetic material know as Pro Osteon Implant 500R. This naturally derived material is made from a non-decorative form of coral, which is subject to a patented thermal process, which converts the coral to hydroxyapatite. Following the conversion the material is no longer coral but a composite of highly resorbable calcium carbonate with a slower resorbing outer layer of calcium phosphate. The material retains the porous, interconnected architecture of coral which gives it a similar structure to cancellous bone, which provides a pathway for bony ingrowth. Allogenix Plus is osteoinductive, serves as a scaffold that will provide the framework necessary for bone growth, and osteoconductive, able to induce bone formation when placed into a site were bone may not normally grow. It has been approved for use in filling craniofacial defects and craniotomies that are no larger than 25 cm2.

Material and Methods: In this study we will recruit 5 subjects of 18 months or older with metopic craniosynostosis who will receive Allogenix Plus and bone dust to fill in small calvarial gaps and compare them to a historical cohort that only received bone dust. The parents of new patients seen in clinic will be asked to participate on a voluntary basis until 5 subjects with of 18 months or older with metopic craniosynostosis undergoing fronto-orbital advancement and cranial vault remodeling have been recruited. They will be advised as to the risks and benefits of the study. Once informed consent has been obtained the patient's will undergo surgery. During surgery the calvarial defects less than 25 cm2 will be measured and filled in with a quantified amount of bone dust and a quantified amount of Allogenix Plus. Pictures will be taken of the different stages of the procedure as is currently standard of care. Once we are done with surgery the patient will obtain a Head CT scan in the immediate post-operative period, as is current standard of care. The patient will then receive our standard post-operative care. During clinic visits at 1 week, 3 weeks, 6 weeks, 12 weeks, 6 months, and 1 year we will evaluate for any potential complications including infection, rejection of transplanted material, and wound breakdown. One year after surgery the patient will undergo another CT of the Head. In this CT scan we will evaluate for bone formation, bone resorption, and bony gaps present. We will then obtain a historical cohort comprised of 5 patients that are age and sex matched to our 5 subjects who received Allogenix Plus by performing a chart review. We will compare through pictures, immediate post-operative CT scans of the Head, and 1 year post-operative CT scans of the Head the defect size and the and percent of ossification of defects with bone dust alone, which is our current standard of care, versus bone dust with Allogenix Plus.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 18 months and 36 months with metopic craniosynostosis undergoing cranial vault remodeling with defects 25 cm squared or less

Exclusion Criteria:

* Allergic reaction to any of the components of the bone substitute Allogenic Plus.

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Percentage of ossification | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Muzaffar, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital and Clinics, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No